CLINICAL TRIAL: NCT06399458
Title: The Relationship Between Primary Lymphedema and Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: feyzabegoglu
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lymphedema of Upper Limb
Keywords: primary lymphedema, hyper mobility, Beighton score
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. group: Patients with lymphedema in the lower extremity
  Interventions: Diagnostic Test: For hypermobility; Beighton score and Brighton revised 1998 Criteria
- 2. group: Patients with lymphedema or no edema in the lower extremities
  Interventions: Diagnostic Test: For hypermobility; Beighton score and Brighton revised 1998 Criteria

INTERVENTIONS:
Diagnostic Test: For hypermobility; Beighton score and Brighton revised 1998 Criteria — Beighton score and Brighton revised 1998 Criteria

SUMMARY:
Lymphoedema is the swelling of one or several parts of the body owing to lymph accumulation in the extracellular space. It is often chronic, worsens if untreated, predisposes to infections and causes an important reduction in quality of life.Primary lymphoedema (PLE) is thought to result from abnormal development and/or functioning of the lymphatic system, can present in isolation or as part of a syndrome, and can be present at birth or develop later in life.

Joint hypermobility ( JH) is a clinical condition characterized an excess range of motion in a joint beyond the physiological range of motion .

It is termed generalized joint hypermobilty (GJH) , when the condition is asymptomatic; when it is associated with symptoms such as arthralgia, soft tissue damage, and joint instability, it is referred to as benign joint hypermobility syndrome (BJHS) .An increase in the proportion of collagen or collagen subtypes, such as type III/type I has been detected in JH . This abnormal collagen structure causes joint laxity, and fragility of the connective tissue increases.

The lymphatic system begins to develop at the end of the fifth gestational week. Lymphatic vessels and lymph nodes develop from the mesoderm. Mesoderm differentiates to form many tissues and structures, including connective tissue, muscle, bone, urogenital and circulatory systems. The relationships between systems developing from the same mesoderm-derived structures (such as carpal tunnel hypermobility, lumbar disc herniation hypermobility, shoulder impigment and adhesive capsulitis hypermobility) and joint hypermobility were examined. There are studies showing that hypermobility may pose a risk for venous insufficiency. In addition, one of the criteria for benign joint hypermobility syndrome is the presence of varicose veins. It has been revealed that the lymphatic system develops embryonicly from the cardinal vein, intersomatic vein and lymphangioblasts. Therefore, the lymphatic system can be considered as a branch of the developmental venous system with endothelial vascular walls. We aimed to investigate the relationship between primary lymphedema and joint hypermobility, as it has not been investigated before in the literature and based on this developmental similarity.

DETAILED DESCRIPTION:
The number of samples for our study was determined as minimum n: 29 people for each group as a result of Power analysis using the GPower program. The number of volunteers we will include in our study is 58, including the primary lymphedema group and the control group with similar characteristics and no lymphedema disease. Patients who have previously come to the lymphedema outpatient clinic due to swelling in their legs and who have been diagnosed with primary lymphedema as a result of the examinations and tests will be included (patients with swelling in their lower extremities, regardless of whether there is an initiating factor, stemmer test+, gode+/-, doppler USG: normal, etiology-oriented; abdominal, inguinal USG patients whose results were normal but whose lymphoscintigraphy showed findings of lymphatic insufficiency). Patients will be called and their joint range of motion will be examined for the Beighton score and the Brighton criteria will be questioned. Male and female patients between the ages of 18-65 with primary lymphedema in their lower extremities and healthy volunteers in the same age range who do not have complaints such as edema or lymphedema in their lower extremities will be included in our study.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with primary lymphedema between the ages of 18-65. Individuals between the ages of 18-65 without a diagnosis of lymphedema. Lymphedema stage 1,2,3 patients. Sufficient cognitive functions.

Exclusion Criteria:

Being diagnosed with secondary lymphedema. Patients with lower extremity edema due to other reasons (such as cardiac, nephrogenic, myxedema), in this context, patients with cardiac failure, renal failure, thyroid hormone disorders Patients using edema-inducing drugs (corticosteroids, calcium channel blockers, gabapentin, pregabalin Patients diagnosed with rheumatological disease Patients with signs of infection in their legs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study included male and female patients between the ages of 18-65 with primary lymphedema in the lower extremities and healthy volunteers in the same age range who did not have complaints such as edema or lymphedema in the lower extremities.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Beighton Hypermobility Score | 1 day
  The following examinations are performed for the Beighton hypermobility score:1. Ability to touch palms flat to floor with knees straight (one point) 2. Elbow extension >10° (one point for each side) 3. Knee extension >10° (one point for each side) 4. Ability to touch thumb to forearm (one point for each side) 5. Fifth finger metocarpalphalageal joint extension >90° (one point for each side) Scores of 4 or above indicate Generalised Joint Hypermobility.
Revised Brighton Criteria | 1 day
  The Brighton Criteria is used in adults to diagnose Joint Hypermobility Syndrome. To make the diagnosis you need one of: two major criteria; one major and two minor criteria; four minor criteria; two minor criteria and one affected first degree relative. The presence of an underlying syndrome excludes the diagnosis.
  Major Criteria:
  Beighton Score >3, Arthralgia > 3 months in four or more joints.
  Minor Criteria:
  Beighton Score 1-3, Arthralgia > 3 months in one joint, backpain, or spondylosis / spondylolysis / ,spondylolisthesis.
  Dislocation or subluxation in more than one joint, or in one joint repeatedly. Three or more soft tissue lesions (e.g epicondylitis, tenosynovitis, bursitis). Marfanoid habitus. Skin striae. Ocular signs (e.g drooping eyelids, myopia, antimongoloid slant). Varicose veins, hernia, uterine or rectal prolapse. Mitral valve prolapse.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Akan Begoğlu, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No